CLINICAL TRIAL: NCT05448144
Title: Alterations of Gut Microbiota and Metabolites in Asian Patients With Alcohol-associated Liver Disease
Brief Title: Alterations of Gut Microbiota and Metabolites in ALD Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Huikuan Chu, MD, Associate chief physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: UHCT22032
Record Dates: First submitted 2022-07-02; First posted 2022-07-07 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Liver Disease; Alcohol-Related; Gut Microbiota
Keywords: Alcohol-associated liver disease; Gut microbiota; Metabonomics
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Retain patient blood and stool and extract DNA for identification of gut microbiota.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Alcohol-associated liver disease: drinking, had fatty liver, hepatitis, or hepatic cirrhosis
  Interventions: Other: Collect stool and blood samples from patients
- Purely drinking: drinking, but had no fatty liver and hepatitis.
  Interventions: Other: Collect stool and blood samples from patients
- Healthy control: no drinking and no liver diseases.
  Interventions: Other: Collect stool and blood samples from patients

INTERVENTIONS:
Other: Collect stool and blood samples from patients — Collect stool and blood samples from patients

SUMMARY:
Alcohol-associated liver disease is one of the most prevalent liver diseases worldwide, and the leading cause of liver transplantation in the U.S. Alcohol-related liver disease is associated with changes in the intestinal microbiota and metabolites.

DETAILED DESCRIPTION:
Backgrounds:

Alcohol-associated liver disease (ALD) is a common disease caused by alcohol use disorder (AUD), ranging from asymptomatic liver steatosis to alcohol-associated hepatitis (AH), alcoholic cirrhosis and potentially, hepatocellular carcinoma (HCC). ALD is the most common reason for liver transplantation in the United States. Globally, about 2 million people die from liver disease each year and up to 50% of the death with cirrhosis can be attributed to alcohol consumption. In Europe, it has been estimated that 60%-80% of liver-related deaths can be attributed to alcohol consumption. Currently, the pathogenetic mechanisms have not been fully elucidated, but they might be related to oxidative stress, acetaldehyde-induced toxicity, cytokine and chemokine-induced inflammation. There is no effective therapeutic method for ALD till now except for liver transplantation. Recent studies have reported that gut microbiota has an intimate relationship with ALD, which provides broader insights and opportunities for understanding and treating this disease.

Aims:

We aim to map the alterations of gut microbiota and metabolites in patients with different levels of ALD, and to investigate the effects and mechanisms of key strains and their metabolites on the development of ALD, providing a theoretical basis and potential targets for its treatment.

Methods:

Patients who meet the inclusion criteria will sign informed consent, their demographic data, clinical labs, serum, and feces for shotgun metagenomics will be collected at baseline.

Anticipated Results:

Compared to healthy control group, patients with AH or alcohol-associated hepatic cirrhosis will suffer from microbiota dysbiosis and have more microbes and microbial genes associated with inflammation and fibrosis. Gut microbiota-derived metabolites may exacerbate the severity of ALD. Several microorganisms or metabolites can be used as prognostic markers.

Implications and Future Studies:

Results of altered gut microbiome and metabolites could provide potential targets for manipulating intestinal microbiota to prevent or treat ALD.

ELIGIBILITY:
Inclusion Criteria:

1. The group of ALD:

1. aged >18 years;
2. patients who meet the diagnostic criteria of ALD in Chinese Guideline for the Prevention and Management of Alcoholic Liver Disease (2018 Update);
3. history of chronic heavy alcohol consumption;
4. with relatively complete clinical data and good compliance.

2. The group of purely drinking:

1. aged >18 years;
2. history of chronic alcohol consumption;
3. no evidence of fatty liver, hepatitis or liver injury.

3. The group of healthy control:

1. aged >18 years;
2. without history of alcohol consumption;
3. no evidence of fatty liver, hepatitis or liver injury.

Exclusion Criteria:

1. with hepatocellular carcinoma or hepatic metastases;
2. combined with infectious liver diseases, such as hepatitis A virus, hepatitis B virus, hepatitis C virus, hepatitis D virus, hepatitis E virus and human immunodeficiency virus (HIV);
3. combined with non-infectious liver diseases, such as non-alcoholic fatty liver disease, drug-induced hepatitis, autoimmune liver disease, Immunoglobulin G subclass 4-related liver disease, Wilson's disease, alpha 1-antitrypsin deficiency, Budd-Chiari syndrome, and other congenital liver diseases;
4. combined with severe organic lesions of other organs;
5. pregnant and lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and healthy control will be recruited mainly from the outpatient or inpatient departments of Wuhan Union Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The alterations of gut microbiota in different groups | When subjects are enrolled
  The alterations will be detected by genome sequencing
The alterations of gut metabolites in different group | When subjects are enrolled
  The alterations will be detected by metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Huikuan Chu, M.D., Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Result] Chu H, Duan Y, Lang S, Jiang L, Wang Y, Llorente C, Liu J, Mogavero S, Bosques-Padilla F, Abraldes JG, Vargas V, Tu XM, Yang L, Hou X, Hube B, Starkel P, Schnabl B. The Candida albicans exotoxin candidalysin promotes alcohol-associated liver disease. J Hepatol. 2020 Mar;72(3):391-400. doi: 10.1016/j.jhep.2019.09.029. Epub 2019 Oct 10. PMID 31606552
- [Result] Duan Y, Llorente C, Lang S, Brandl K, Chu H, Jiang L, White RC, Clarke TH, Nguyen K, Torralba M, Shao Y, Liu J, Hernandez-Morales A, Lessor L, Rahman IR, Miyamoto Y, Ly M, Gao B, Sun W, Kiesel R, Hutmacher F, Lee S, Ventura-Cots M, Bosques-Padilla F, Verna EC, Abraldes JG, Brown RS Jr, Vargas V, Altamirano J, Caballeria J, Shawcross DL, Ho SB, Louvet A, Lucey MR, Mathurin P, Garcia-Tsao G, Bataller R, Tu XM, Eckmann L, van der Donk WA, Young R, Lawley TD, Starkel P, Pride D, Fouts DE, Schnabl B. Bacteriophage targeting of gut bacterium attenuates alcoholic liver disease. Nature. 2019 Nov;575(7783):505-511. doi: 10.1038/s41586-019-1742-x. Epub 2019 Nov 13. PMID 31723265
- [Result] Chu H, Duan Y, Yang L, Schnabl B. Small metabolites, possible big changes: a microbiota-centered view of non-alcoholic fatty liver disease. Gut. 2019 Feb;68(2):359-370. doi: 10.1136/gutjnl-2018-316307. Epub 2018 Aug 31. PMID 30171065
- [Result] Jiang L, Chu H, Gao B, Lang S, Wang Y, Duan Y, Schnabl B. Transcriptomic Profiling Identifies Novel Hepatic and Intestinal Genes Following Chronic Plus Binge Ethanol Feeding in Mice. Dig Dis Sci. 2020 Dec;65(12):3592-3604. doi: 10.1007/s10620-020-06461-6. Epub 2020 Jul 15. PMID 32671585
- [Result] Chu H, Williams B, Schnabl B. Gut microbiota, fatty liver disease, and hepatocellular carcinoma. Liver Res. 2018 Mar;2(1):43-51. doi: 10.1016/j.livres.2017.11.005. Epub 2018 Feb 21. PMID 30416839
- See also: This web provides information of Human Subjects Protection in this study — https://gcp.whuh.com/index.aspx

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT05448144/Prot_SAP_ICF_000.pdf